CLINICAL TRIAL: NCT03519919
Title: Clariti 1-Day Multifocal Study - 'Real World' Subjective Acceptance Study (HARP)
Brief Title: Somofilcon A 1-Day Multifocal Study - Real World Subjective Acceptance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-MKTG-81
Record Dates: First submitted 2018-05-01; First posted 2018-05-09 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Somofilcon A multifocal lens (Experimental): Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment.
  Interventions: Device: somofilcon A multifocal lens

INTERVENTIONS:
Device: somofilcon A multifocal lens — contact lens
  Other Names: clarifi multifocal lens

SUMMARY:
The objective of the study is to evaluate the performance of somofilcon A 1 day multifocal when worn on a daily disposable wear modality over a period of up to 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Has had a self-reported oculo-visual examination in the last two years.
* Currently wears multifocal soft contact lenses, and have worn multifocal contact lenses for at least one month;
* Presently wears lenses for minimum wear 4 days/week and 10 hours/day
* Participant has an anticipated ability to wear test lenses for minimum 5 days/week and 10 hours/day.
* Can be fit with the available test contact lens power range to achieve satisfactory vision i.e. 0.18 logMar (20/30) binocular distance acuity with the test lenses.
* Current refraction indicates a reading addition of +1.50 or higher
* Uses a digital device (computer/laptop/tablet etc.) for at least 5hrs/day
* Spends 10 hrs or more indoors at least 5 days/week
* Possesses a smartphone and is willing to download the MetricWire app to receive

Exclusion Criteria:

* Is presently wearing Clariti 1 day multifocal lenses
* Has astigmatism greater than -0.75 DCyl as determined with subjective refraction
* Is participating in any concurrent clinical or research study;
* Has any known active* ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to fluorescein dye or products to be used in the study;
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
* Is aphakic;
* Has undergone refractive error surgery;
* Is an employee of the Centre for Contact Lens Research

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Somofilcon A Multifocal Lens
Started | 51
Completed | 48
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Population: Fifty-one participants were enrolled in the study. Habitual wearers of multifocal soft contact lenses were refit with clariti 1day multifocal. 48 participants completed the study.
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Vision Clarity During the Day - Distance Vision
Description: Subjective expectation -Vision clarity during the day - distance vision was measured from three subjective expectation responses completed at the office. The responses were assigned numbers as below:
  Fell short of expectations = 1 Met my expectations = 2 Exceeded my expectations = 3
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Habitual Lens -Distance Vision While Driving During the Day; Habitual Lens - Distance Tasks in Good Lighting.; Habitual Lens - Distance Tasks in General: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment.
  Contact Lens: Habitual Lens
Arm/Group | Habitual Lens -Distance Vision While Driving During the Day | Habitual Lens - Distance Tasks in Good Lighting. | Habitual Lens - Distance Tasks in General
Number analyzed (Participants) | 48 | 48 | 48
percentage of participants
  Fell short of my expectations | 22.9 | 14.6 | 27.1
  Met my expectations | 68.8 | 77.1 | 68.7
  Exceeded my expectations | 8.3 | 8.3 | 4.2

2. Primary Outcome: Vision Clarity During the Day - Distance Vision
Description: Subjective expectation - Vision clarity during the day - distance vision was measured from three subjective expectation responses completed at the office. The responses were assigned numbers as below:
  Fell short of expectations = 1 Met my expectations = 2 Exceeded my expectations = 3
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Groups:
- Somofilcon A Multifocal Lens - Distance Vision While Driving: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment..
  Contact lens : somofilcon A multifocal lens
- Somofilcon A Multifocal Lens -Distance Tasks in Good Lighting; Somofilcon A Multifocal Lens-Distance Tasks in General: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment.
  Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens - Distance Vision While Driving | Somofilcon A Multifocal Lens -Distance Tasks in Good Lighting | Somofilcon A Multifocal Lens-Distance Tasks in General
Number analyzed (Participants) | 48 | 48 | 48
percentage of participants
  Fell short of my expectations | 16.7 | 12.5 | 18.8
  Met my expectations | 64.5 | 70.8 | 64.5
  Exceeded my expectations | 18.8 | 16.7 | 16.7

3. Secondary Outcome: Number of Participants With Lens Centration
Description: Lens centration on the cornea (Optimum, Acceptable decentration, Unacceptable decentration (>=0.5mm))
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Lens Centration at baseline.
  Contact Lens: Habitual Lens
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Lens Centration at baseline.
  Contact lens : somofilcon A multifocal lens
Arm/Group | Habitual Lens | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48 | 48
Participants
  Optimum | 40 | 34
  Acceptable decentration | 8 | 14
  Unacceptable decentration | 0 | 0

4. Secondary Outcome: Number of Participants With Lens Centration
Description: Lens centration on the cornea (Optimum, Acceptable decentration, Unacceptable decentration (>=0.5mm))
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Lens Centration Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
Participants
  Optimum | 32
  Acceptable decentration | 16
  Unacceptable decentration | 0

5. Secondary Outcome: Visual Acuity
Description: Distance visual acuity (logMAR)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: logMar
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and - Lens Centration at baseline.
  Contact Lens: Habitual Lens
Arm/Group | Habitual Lens | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48 | 48
logMar
  Right Eye | 0.10 (0.12) | 0.02 (0.11)
  Both Eyes | -0.01 (0.09) | -0.05 (0.08)

6. Secondary Outcome: Visual Acuity
Description: Distance visual acuity (logMAR)
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: logMar
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and - Visual Acuity Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
logMar
  Right Eye | 0.00 (0.09)
  Both Eyes | -0.04 (0.09)

7. Secondary Outcome: Post-blink Lens Movement
Description: Movement of lens on eye after blink was graded on a 5-point Likert scale (0-4, 1 steps) as follows: 0 - insufficient, 1 - minimal but acceptable, 2 - optimal, 3 - moderate but acceptable, and 4 - excessive unacceptable movement.
Time Frame: Baseline
Measure: Number; unit: percentage of particpants
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Post blink movement at baseline.
  Contact Lens: Habitual Lens
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Post blink movement at baseline.
  Contact lens : somofilcon A multifocal lens
Arm/Group | Habitual Lens | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48 | 48
percentage of particpants
  Insufficient | 0 | 0
  Minimal, but acceptable movement | 20.8 | 8.3
  Optimal Movement | 72.9 | 70.8
  Moderate, but acceptable Movement | 6.3 | 20.8
  Excessive unacceptable | 0 | 0

8. Secondary Outcome: Post-blink Lens Movement
Description: Movement of lens on eye after blink was graded on a 5-point scale (0-4, 1 steps) as follows: 0 - insufficient, 1 - minimal but acceptable, 2 - optimal, 3 - moderate but acceptable , and 4 - excessive unacceptable.
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment - Post blink movement
  Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Insufficient | 0
  Minimal, but acceptable movement | 8.3
  Optimal Movement | 77.1
  Moderate, but acceptable Movement | 14.6
  Excessive unacceptable | 0

9. Secondary Outcome: Corneal Staining
Description: Corneal staining will be assessed for extent (0-100) with 0 indicating no staining/indentation and 100 indicating deep confluent staining or severe indentation for following regions: Temporal, Superior, Nasal, Inferior and Central.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Corneal Staining at Baseline.
  Contact Lens: Habitual Lens
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
units on a scale
  Temporal | 1.15 (4.28)
  Superior | 1.15 (4.28)
  Nasal | 1.35 (5.03)
  Inferior | 2.81 (6.60)
  Central | 1.88 (6.87)

10. Secondary Outcome: Corneal Staining
Description: as for outcome 9
Time Frame: 3 weeks
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and - corneal staining Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
units on a scale
  Temporal | 1.77 (7.75)
  Superior | 1.04 (3.57)
  Nasal | 1.15 (4.03)
  Inferior | 3.06 (9.54)
  Central | 0.75 (3.57)

11. Secondary Outcome: Conjunctival Staining
Description: Conjunctival staining will be assessed using CORE integer scale (0-100) with 0 indicating no staining/indentation and 100 indicating deep confluent staining or severe indentation for following regions: Temporal, Superior, Nasal, Inferior.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Conjunctival Staining at Baseline.
  Contact Lens: Habitual Lens
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
units on a scale
  Temporal | 10.31 (12.3)
  Superior | 7.70 (12.8)
  Nasal | 11.04 (13.0)
  Inferior | 9.69 (13.0)

12. Secondary Outcome: Conjunctival Staining
Description: Conjunctival staining will be assessed using CORE integer scale (0-100) with 0 indicating no staining/indentation and 100 indicating deep confluent staining or severe indentationfor following regions: Temporal, Superior, Nasal, Inferior.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - conjunctival staining Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
units on a scale
  Temporal | 16.87 (22.2)
  Superior | 7.60 (15.0)
  Nasal | 12.7 (17.2)
  Inferior | 11.8 (19.5)

13. Secondary Outcome: Bulbar Hyperemia
Description: Grading hyperemia of bulbar conjunctiva on a scale ranged from 0-4 and in 0.50 steps, with 0 indicating no hyperemia and 4 indicating severe hyperemia.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - Bulbar hyperemia at Baseline.
  Contact Lens: Habitual Lens
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
units on a scale
  Bulbar Hyperemia | 2.10 (0.65)
  Limbal Hyperemia | 1.90 (0.69)

14. Secondary Outcome: Bulbar Hyperemia
Description: as for outcome 13
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens - bulbar hyperemia Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
units on a scale
  Bulbar Hyperemia | 2.05 (0.57)
  Limbal Hyperemia | 1.90 (0.71)

15. Secondary Outcome: Subjective Vision Satisfaction - Driving at Night
Description: Subjective satisfaction of distance vision while driving at night responses for habitual lens (1= fell short of expectation, 2 = met expectation, 3= exceed expectation)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment.
  Contact Lens: Habitual Lens
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 22.9
  Met expectations | 68.8
  Exceeded expectations | 8.3

16. Secondary Outcome: Subjective Vision Satisfaction - Driving at Night
Description: Subjective satisfaction of distance vision while driving at night responses for somofilcon A multifocal lens (1= fell short of expectation, 2 = met expectation, 3= exceed expectation)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment.
  Contact lens : somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 16.7
  Met expectations | 64.6
  Exceeded expectations | 18.8

17. Secondary Outcome: Subjective Vision Satisfaction - Long Intermediate Vision
Description: Subjective satisfaction of long intermediate vision while using desktop computer for habitual lens (1= fell short of expectation, 2= met expectation, 3= exceed expectation)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 12.5
  Met expectations | 85.4
  Exceeded expectation | 2.1

18. Secondary Outcome: Subjective Vision Satisfaction - Long Intermediate Vision
Description: Subjective satisfaction of long intermediate vision while using desktop computer for somofilcon A multifocal lens (1= fell short of expectation, 2= met expectation, 3= exceed expectation)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment.
  Contact Lens: somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 8.3
  Met expectations | 66.7
  Exceeded expectation | 25.0

19. Secondary Outcome: Subjective Vision Satisfaction - Short Intermediate Tasks
Description: Subjective satisfaction of short/intermediate vision while using laptop/tablet for habitual lens (1= fell short of expectation, 2= met expectation, 3= exceed expectation)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 22.9
  Met expectations | 70.8
  Exceeded expectations | 6.3

20. Secondary Outcome: Subjective Vision Satisfaction - Short Intermediate Tasks
Description: Subjective satisfaction of short/intermediate vision while using laptop/tablet for somofilcon A multifocal lens (1= fell short of expectation, 2= met expectation, 3= exceed expectation)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 14.6
  Met expectations | 62.5
  Exceeded expectations | 22.9

21. Secondary Outcome: Subjective Vision Satisfaction - Near Vision
Description: Subjective satisfaction of near vision while reading on cell phone and hand-held materials for habitual lens (1 = fell short of expectation, 2 = met expectation, 3 = exceed expectation)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 43.8
  Met expectations | 50.0
  Exceeded expectations | 6.2

22. Secondary Outcome: Subjective Vision Satisfaction - Near Vision
Description: Subjective satisfaction of near vision while reading on cell phone and hand-held materials for somofilcon A multifocal lens (1 = fell short of expectation, 2 = met expectation, 3 = exceed expectation)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Groups:
- Somofilcon A Multifocal Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment.
  Contact Lens:somofilcon A multifocal lens
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 16.7
  Met expectations | 56.3
  Exceeded expectations | 27.0

23. Secondary Outcome: Ease of Insertion
Description: Subjective rating how easy lens was inserted on eye for habitual lens (1 = Fell short of expectation, 2 = Met expectation, 3 = Exceeded expectations)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Habitual Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment
  Contact Lens: Habitual Lens
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 6.3
  Met expectations | 81.3
  Exceeded expectations | 12.4

24. Secondary Outcome: Ease of Insertion
Description: Subjective rating how easy lens was inserted on eye for somofilcon A multifocal lens (1 = Fell short of expectation, 2 = Met expectation, 3 = Exceeded expectations)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 6.3
  Met expectations | 60.4
  Exceeded expectations | 33.3

25. Secondary Outcome: Ease of Removal
Description: Subjective rating for habitual lens on how easy lens was removed from eye (1 = Fell short of expectation, 2 = Met expectation, 3 = Exceeded expectations)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 4.2
  Met expectations | 83.3
  Exceeded expectations | 12.5

26. Secondary Outcome: Ease of Removal
Description: Subjective rating for somofilcon A multifocal lens on how easy lens was removed from eye (1 = Fell short of expectation, 2 = Met expectation, 3 = Exceeded expectations)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 14.6
  Met expectations | 62.5
  Exceeded expectations | 22.9

27. Secondary Outcome: Overall Satisfaction With Speed of Changing Focus
Description: Subjective rating for speed and ability to change focus between distances for habitual lens (1 = Fell short of expectation, 2 = Met expectation, 3 = Exceeded expectations)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 12.5
  Met expectations | 75.0
  Exceeded expectations | 12.5

28. Secondary Outcome: Overall Satisfaction With Speed of Changing Focus
Description: Subjective rating for speed and ability to change focus between distances for somofilcon A multifocal lens (1 = Fell short of expectation, 2 = Met expectation, 3 = Exceeded expectations)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell short of expectations | 6.3
  Met expectations | 66.7
  Exceeded expectations | 27.0

29. Secondary Outcome: Overall Satisfaction Preference Between Study and Habitual Contact Lenses
Description: Subjective satisfaction preference of contact lens between study and habitual contact lenses(Fell short of expectations, Met my expectation, Exceeded my expectation)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell Short of expectations | 18.8
  Met expectations | 68.8
  Exceeded expectations | 12.4

30. Secondary Outcome: Overall Satisfaction Preference Between Study and Habitual Contact Lenses
Description: Subjective satisfaction preference between study and habitual contact lenses (Fell short of expectations, Met ,my expectations, Exceeded my expectations))
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A Multifocal Lens
Number analyzed (Participants) | 48
percentage of participants
  Fell Short of expectations | 14.6
  Met expectations | 58.3
  Exceeded expectations | 27.1

31. Secondary Outcome: Overall Comfort
Description: Subjective rating of comfort for habitual lens and somofilcon A multifocal lens at 3 weeks (Prefer my own strongly, Prefer my own slightly, No preference, Prefer study lenses slightly, Prefer study lenses strongly)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Groups:
- Overall Participants: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment at the final visit for overall comfort.
  Contact Lens: somofilcon A 1-day multifocal Contact Lens: Habitual Lens
Arm/Group | Overall Participants
Number analyzed (Participants) | 48
percentage of participants
  Prefer my own strongly | 14.6
  Prefer my own slightly | 10.4
  No preference | 22.9
  Prefer study lenses slightly | 14.6
  Prefer study lenses strongly | 37.5

32. Secondary Outcome: Overall Preference Between Study and Habitual Contact Lenses for Lifestyle
Description: Preference of contact lens for the whole range of tasks (Prefer strongly, Prefer slightly, No preference, Prefer study lenses slightly, Prefer study lenses strongly)
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Groups:
- Overall Study -Do You Prefer Your Own Lenses or the Study Lens: Habitual wearers of multifocal contact lenses will be refit to somofilcon A multifocal lens and provide a subjective assessment at the final visit for overall preference.
  Contact lens - Habitual Lens and somofilcon A contact lens
Arm/Group | Overall Study -Do You Prefer Your Own Lenses or the Study Lens
Number analyzed (Participants) | 48
percentage of participants
  Prefer my own strongly | 14.5
  Prefer my own slightly | 14.6
  No Preference | 18.8
  Prefer study lenses slightly | 22.9
  Prefer study lenses strongly | 29.2

ADVERSE EVENTS:
Time Frame: From baseline visit of habitual lens through follow up visit of somofilcon A multifocal lens for an average of 3 weeks
Arm/Group | Somofilcon A Multifocal Lens
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03519919/Prot_SAP_000.pdf